CLINICAL TRIAL: NCT01394042
Title: Exploratory Evaluation of a Transrectal Scintigraphic Detector (Proxiscan) for Detection of Primary Prostate Cancer Utilizing a Radiotracer Targeting Prostate Specific Membrane Antigen (PMSA)
Brief Title: Prostate Cancer Imaging With Radioactive Tracer and Ultrasound Detector Compared to MRI and ProstaScint
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Radiological Associates of Sacramento Medical Group Inc. (Other)
Collaborators: Hybridyne Imaging Technologies (Unknown)
Responsible Party: Benjamin Franc, MD/PI, RAS
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: Proxiscan
Record Dates: First submitted 2011-07-01; First posted 2011-07-14 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Prostate Cancer
Keywords: Biopsy proven primary prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No intervention (No Intervention): All consenting patients will be imaged with the Proxiscan and data compared with MRI, ProstaScint and biopsy data
  Interventions: Device: Proxiscan device

INTERVENTIONS:
Device: Proxiscan device — All patients will be imaged with the device

SUMMARY:
This is a small study to determine if probe, similar to an ultrasound probe, can detect prostate cancer more specifically than other imaging studies in patients with a positive prostate cancer biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Primary prostate cancer proven by sextant prostate biopsy
* Transrectal ultrasound (TRUS)-guided prostate biopsy within 6 months of study enrollment
* Sufficient time period to complete imaging protocol and 5-7 day safety followup assessment without other therapeutic intervention
* In the judgement of principal investigator, patient able to provide informed consent and be compliant with protocol requirements
* ECOG status of 0 or 1 Pt > 18 yrs of age

Exclusion Criteria:

* Definitive or concomitant therapeutic intervention within the interval of study intervention
* Prior pelvic therapeutic radiation
* Active malignancy or therapy for malignancy with 6 months other than basal or squamous cell carcinoma of the skin
* Pt received radiopharmaceutical which was within 5 half-lives at the time of studying imaging
* Known history of human-anti-murine-antibodies or known allergic reaction to previously received murine based products

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Detection of PSMA antibody (ProstaScint)uptake patterns measured by Proxiscan in comparison with anatomic biopsy reports, conventional SPECT and MRI scans within one month of Proxiscan | Within on month of scan and corresponding MRI
  Detection of PSMA antibody (ProstaScint) uptake patterns measured by the new transrectal compact gamma camera (Proxiscan) will be compared to the anatomic biopsy reports along with Magnetic Resonance Imaging (MRI) and conventional ProstaScint (Single Photon Emission Computed Tomography) SPECT imaging results. All imaging and biopsy results performed within one month will be used for this investigation

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Franc, MD, Principal Investigator — Radiological Associates of Sacramento Medical Group Inc.
Locations (1):
- Roseville PET and Nuclear Imaging Center, Roseville, California, United States